CLINICAL TRIAL: NCT05931445
Title: Multicenter, Open-label, Randomized, Controlled Study to Test the Utility of Electronic Patient-reported Outcome (ePRO) Monitoring in Patients With Unresectable Advanced Cancers or Metastatic/Recurrent Solid Tumors
Brief Title: Patient Reported Outcomes Study Using Electronic Monitoring System for Advanced or Metastatic Solid Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comprehensive Support Project for Oncology Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-MOTE
Record Dates: First submitted 2023-06-05; First posted 2023-07-05 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Lung Cancer; Colorectal Cancer; Liver Cancer; Stomach Cancer; Endometrial Cancer; Ovarian Cancer; Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Liver Neoplasms; Stomach Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring group (Experimental): ePRO monitoring will be conducted once weekly after study enrollment, along with standard care of treatment.
  Interventions: Other: e-PRO monitoring
- Non-monitoring group (No Intervention): Standard care of treatment will be given without ePRO monitoring.

INTERVENTIONS:
Other: e-PRO monitoring — The e-PRO monitoring will concern treatment of each predefined type of cancer or characteristic symptoms of the condition. PRO-CTCAE (Patient-Reported Outcome-Common Terminology Criteria for Adverse Events) will be used as the scale for monitoring symptoms. The patient and (sub)investigator will share the monitoring results during examinations and use them to determine treatment strategies, etc. Threshold values will be predefined for a diagnosis of "severe" for individual symptoms. When it is reported that a threshold value has been exceeded, an alert notification will be sent to the study staff member assigned to the patient. The (sub)investigator who receives the notification will assess the information in the notification and take the best course of action.
  Arms: Monitoring group

SUMMARY:
This is a multicenter, open-label, randomized, controlled study to test the hypothesis that ePRO monitoring added to usual care helps prolong OS or maintain and improve HRQoL in patients with unresectable advanced cancers or metastatic/recurrent solid tumors receiving systemic drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable, advanced, metastasized, or relapsed solid tumors (Breast Cancer, Lung Cancer, Colorectal Cancer, Liver Cancer, Stomach Cancer, Endometrial Cancer, Ovarian Cancer, or Squamous Cell Carcinoma of the Head and Neck)
2. Expected to be able to undergo treatment or observation for at least 6 months at the study site
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1, or 2
4. Receiving systemic anticancer mono- or combination pharmacotherapy (e.g., cytotoxic anticancer agents, molecularly targeted drugs, and immune checkpoint inhibitors) at enrollment or scheduled to begin such therapy within 1 month from the date of enrollment (In principle, patients should be receiving pharmacotherapy on an out-patient basis.)
5. Capable of using electronic device (includes cases needing some assistance)
6. Aged 18 years or older at informed consent
7. Written consent for the study personally obtained from the subject

Exclusion Criteria:

1. Has undergone four or more regimens of pharmacotherapy for advanced, metastasized, or relapsed solid tumors*Notes 1, 2
2. Currently participating in a study where PRO is tracked and the results are passed on to a physician
3. The following are exclusion criteria for individual types of cancer 1) Breast cancer

   * Scheduled to receive or currently receiving endocrine therapy (including endocrine therapy in combination with other agents) for hormone receptor-positive breast cancer
   * Scheduled to receive or currently receiving first regimen of anti-HER2 therapy for HER2-positive disease 2) Liver cancer
   * Hepatic function of Child-Pugh B/C
4. Undergoing or scheduled to undergo radiation therapy for curative purposes
5. Deemed otherwise unsuitable for the study by the investigator or sub-investigator

   * Notes:

     1. If the disease has relapsed during perioperative adjuvant chemotherapy or within 24 weeks after adjuvant chemotherapy, the adjuvant chemotherapy will be considered as the first regimen of adjuvant chemotherapy.
     2. Does not include endocrine therapy for breast cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | After enrollment to death from any cause (up to 57 months)
HRQoL EORTC Quality of Life of Cancer Patients (QLQ-C30) global health status score | At enrollment and week 4,8,12,16,20 and 24 after enrollment

SECONDARY OUTCOMES:
HRQoL EORTC Quality of Life of Cancer Patients (QLQ-C30) domain score | At enrollment and week 4,8,12,16,20 and 24 after enrollment
HRQoL EQ-5D-5L index score | At enrollment and every 4 weeks after enrollment up to 57 months
Quality-adjusted life year (QALY) score | After enrollment to death from any cause (up to 57 months)
At-home mortality rate | After enrollment to death from any cause (up to 57 months)
Time from last completion of drug therapy to death | Time from last completion of drug therapy to death from any cause (up to 57 months)
Number of unscheduled hospital visits during drug therapy | After enrollment up to 24 weeks
Relative Dose Intensity (RDI) | After enrollment up to 24 weeks
Total number of drug regiments | After enrollment up to 57 months
Incremental Cost-Effectiveness Ratio (ICER) | After enrollment up to 57 months
Communication between patients and healthcare providers (EORTC QLQ-COMU26 score) | At enrollment and week 24 after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Hironobu Minami, Principal Investigator — Kobe University Graduate School
Locations (1):
- Kobe University Graduate School, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No